CLINICAL TRIAL: NCT06341127
Title: A Single Patient Trial of Fluoxetine in KCNC1-related Disorder
Brief Title: Fluoxetine in KCNC1-related Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01
Record Dates: First submitted 2024-02-12; First posted 2024-04-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: KCNC1 Related Disorder; Genetic Disease; Rare Diseases
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases | interventions — Fluoxetine

STUDY DESIGN:
Masking Description: This quasi experimental design involves masking of transition moments, but the investigator and participant are aware of the order of cross-over.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Placebo-Fluoxetine-Placebo (Experimental): placebo (medical grade cornstarch in a gel capsule, 1 capsule daily), followed by blinded randomized cross-over moment to active fluoxetine (2.5 then 5 mg po daily), followed by blinded randomized cross-over moment back to placebo
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Oral fluoxetine daily, 2.5 to 5 mg.

SUMMARY:
This is a single patient study of oral powdered fluoxetine to target developmental outcomes in a child with KCNC1-related disorder. This trial will be conducted at Holland Bloorview Kids Rehabilitation Hospital over 32 to 42 weeks, using a quasi experimental ABA phase design (placebo-fluoxetine-placebo) with randomized and blinded active treatment start and stop moments.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided by substitute decision maker.
2. In good general health as evidenced by medical history
3. Screening baseline bloodwork (or availability of clinical bloodwork within 3 months of trial start) with values below relevant cut-offs for adequate hepatic and renal function, and baseline electrolytes including potassium within normal range.
4. Ability to take oral medication and be willing to adhere to the daily oral medication regimen

Exclusion Criteria:

1. Current use of monoamine oxidase inhibitors, other selective serotonin reuptake inhibitors, tricyclic antidepressants, or agents that strongly affect metabolism via CYP2D6, CYP2C9 or CYP3A4.
2. Hypersensitivity to fluoxetine or to any ingredient in the formulation, including any non-medicinal ingredient, or component of the container
3. Treatment with another investigational drug or other medication intervention within 8 weeks of starting the trial.
4. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk.
5. Long QT syndrome including acquired long QT syndrome (e.g., due to concomitant use of a drug that prolongs the QT); a family history of QT prolongation; or other clinical conditions that predispose to arrhythmias.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Motor development | Weekly from date of randomization to up to 42 weeks
  Parent report on the Early Motor Questionnaire
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of randomization to up to 42 weeks
  Adverse event reporting

SECONDARY OUTCOMES:
Adaptive skills | Week 1, 13, 29 and 37
  Vineland Adaptive Behavior Scale
Cognitive skills | Week 1, 13, 29 and 37
  Mullen Scales of Early Learning
Family priority outcome targets | Weekly from date of randomization to up to 42 weeks
  Measure Your Own Medical Profile- 2
Clinical Global Impression- Improvement Scale (CGI-I) | Every 4 weeks from date of randomization to up to 42 weeks
  Clinician assessment of overall development

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Baribeau, MD, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Single patient trial; would be challenging to de-identify.